CLINICAL TRIAL: NCT04373876
Title: Experience From the Long-term Italian Subcutaneous Implantable Cardioverter Defibrillator Registry (ELISIR)
Brief Title: Experience From the Italian S-ICD Registry
Acronym: ELISIR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Luigi Sacco University Hospital (Other)
Responsible Party: Principal Investigator, Giovanni B Forleo, Section head electrophysiology and cardiac pacing, Luigi Sacco University Hospital
Other Study IDs: S-ICD-ITA
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Sudden Cardiac Death; Cardiac Arrest; Ventricular Arrythmia; Implantable Cardiac Defibrillator
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Subcutaneous Implantable Cardioverter Defibrillator — Patients implanted with a totally subcutaneous defibrillator system

SUMMARY:
The purpose of this registry is to collect data on implant parameters, early, mid and long-term clinical effectiveness of Subcutaneous Implantable Cardioverter Defibrillator (S-ICD) therapies in order to better understand how to improve the clinical care of patients and effectiveness of S-ICD therapies.

DETAILED DESCRIPTION:
ISIR is an observational, multicentric registry designed to collect implant and follow-up data of consecutive patients implanted with Subcutaneous Implantable Cardioverter Defibrillator (S-ICD).

A number of about 10 enrolling centers is estimated with an overall number of 400 patients.

A minimal follow-up of 6 months is required before analyzing clinical outcomes. The data analysis will focus on implant outcomes and early, mid and long-term effectiveness of S-ICD therapies and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Patients successfully implanted with S-ICD
* Patients able to provide written informed consent or have informed consent as provided by a legal representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with S-ICD implanted for primary or secondary prevention of sudden cardiac death
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Mortality | 2 years
  Overall or arrhythmic mortality
Appropriate shocks | 2 years
  Appropriate therapies delivered by the devices
Inappropriate shocks | 2 years
  Inappropriate therapies delivered by the devices

CONTACTS AND LOCATIONS:
Locations (18):
- Pitié-Salpêtrière University Hospital, Paris, France
- Asklepios Klinik St. Georg, Hamburg, Germany
- Italy (15):
  - Azienda Sanitaria Provinciale di Cosenza "Ospedale di Castrovillari", Castrovillari, Cosenza
  - Presidio Ospedaliero Di Anzio e Nettuno, Anzio, Rome
  - Presidio Ospedaliero G. B. Grassi, Lido di Ostia, Rome
  - Presidio Ospedaliero G. Salesi, Ancona
  - Policlinico Sant'Orsola-Malpighi, Bologna
  - Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedale Vito Fazzi, Lecce
  - Centro Cardiologico Monzino, IRCCS, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Ospedale Luigi Sacco - Polo Universitario, Milan
  - Ospedale San Gerardo, Monza
  - Policlinico Universitario Campus Bio-Medico, Rome
  - Ospedale San Filippo Neri, Rome
  - Policlinico Umberto I, Rome
- University Hospital of Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gulletta S, Gasperetti A, Schiavone M, Vogler J, Fastenrath F, Breitenstein A, Laredo M, Palmisano P, Mitacchione G, Compagnucci P, Kaiser L, Hakmi S, Angeletti A, De Bonis S, Picarelli F, Arosio R, Casella M, Steffel J, Fierro N, Guarracini F, Santini L, Pignalberi C, Piro A, Lavalle C, Pisano E, Viecca M, Curnis A, Badenco N, Ricciardi D, Dello Russo A, Tondo C, Kuschyk J, Della Bella P, Biffi M, Forleo GB, Tilz R. Age-related differences and associated mid-term outcomes of subcutaneous implantable cardioverter-defibrillators: A propensity-matched analysis from a multicenter European registry. Heart Rhythm. 2022 Jul;19(7):1109-1115. doi: 10.1016/j.hrthm.2022.02.029. Epub 2022 Mar 5. PMID 35257974
- [Derived] Forleo GB, Gasperetti A, Breitenstein A, Laredo M, Schiavone M, Ziacchi M, Vogler J, Ricciardi D, Palmisano P, Piro A, Compagnucci P, Waintraub X, Mitacchione G, Carrassa G, Russo G, De Bonis S, Angeletti A, Bisignani A, Picarelli F, Casella M, Bressi E, Rovaris G, Calo L, Santini L, Pignalberi C, Lavalle C, Viecca M, Pisano E, Olivotto I, Curnis A, Dello Russo A, Tondo C, Love CJ, Di Biase L, Steffel J, Tilz R, Badenco N, Biffi M. Subcutaneous implantable cardioverter-defibrillator and defibrillation testing: A propensity-matched pilot study. Heart Rhythm. 2021 Dec;18(12):2072-2079. doi: 10.1016/j.hrthm.2021.06.1201. Epub 2021 Jun 30. PMID 34214647
- [Derived] Ricciardi D, Ziacchi M, Gasperetti A, Schiavone M, Picarelli F, Diemberger I, Bontempi L, Di Belardino N, Bisignani G, De Bonis S, Mitacchione G, Calabrese V, Lavalle C, Piro A, Pignalberi C, Santini L, Grigioni F, Tondo C, Biffi M, Forleo GB. Clinical impact of defibrillation testing in a real-world S-ICD population: Data from the ELISIR registry. J Cardiovasc Electrophysiol. 2021 Feb;32(2):468-476. doi: 10.1111/jce.14833. Epub 2020 Dec 18. PMID 33296533